CLINICAL TRIAL: NCT07306585
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity Characteristics and Preliminary Efficacy of Multiple Ascending Doses of HC022 Injection in Subjects With Systemic Lupus Erythematosus and/or Cutaneous Lupus Erythematosus
Brief Title: The Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of HC022 Injection in Subjects With SLE/CLE
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HC Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BT-HC022-102
Record Dates: First submitted 2025-09-05; First posted 2025-12-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE); Cutaneous Lupus Erythematosus (CLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HC022 100mg (Experimental): Participants will receive subcutaneous (SC) dose of 100 mg HC022 or matching placebo with a dosing frequency of Q4W (once every 4 weeks), administered subcutaneously twice.
  Interventions: Drug: HC022; Drug: Placebo
- HC022 225mg (Experimental): Participants will receive subcutaneous (SC) dose of 225mg HC022 or matching placebo with a dosing frequency of Q4W (once every 4 weeks), administered subcutaneously twice.
  Interventions: Drug: HC022; Drug: Placebo
- HC022 450mg (Experimental): Participants will receive subcutaneous (SC) dose of 450mg HC022 or matching placebo with a dosing frequency of Q4W (once every 4 weeks), administered subcutaneously twice.
  Interventions: Drug: HC022; Drug: Placebo
- HC022 450mg-2 (Experimental): Participants will receive subcutaneous (SC) dose of 450mg HC022 or matching placebo with a dosing frequency of Q4W (once every 4 weeks),1 additional dose at the end of Week 2 (D15) for a total of 3 doses
  Interventions: Drug: HC022; Drug: Placebo

INTERVENTIONS:
Drug: HC022 — Administered as specified in the treatment arm
Drug: Placebo — Administered as specified in the treatment arm

SUMMARY:
The primary objective of this phase Ib study is to evaluate the safety and tolerability of multiple-ascending, subcutaneous (SC) doses of HC022 in SLE/CLE subjects. Secondary objectives of study are as follows: To estimate the PK parameters of multiple-ascending SC doses of HC022 in SLE/CLE subjects；To evaluate the immunogenicity of HC022 administered to SLE/CLE subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who voluntarily participate in the study, are able to sign the informed consent form and comply with the requirements on the informed consent form;
* 2. Age ≥ 18 years, regardless of gender;
* 3. Subjects and their partners have no birth plan during the study treatment period and within 6 months after the last dose, and voluntarily use effective and reliable contraception (Attachment 1). Female subjects must have a negative serum pregnancy test and be non-lactating;
* 4. Patients diagnosed with SLE or CLE by the investigator

Exclusion Criteria:

* 1. active severe lupus nephritis
* 2. active neuropsychiatric SLE
* 3 .History or current diagnosis of any other systemic autoimmune disease other than secondary Sjogren's syndrome, including but not limited to rheumatoid arthritis, psoriatic arthritis, dermatomyositis, systemic sclerosis (scleroderma), clinically significant non-SLE related vasculitis;
* 4. Drug-induced lupus;
* 5. HIV medical history or positive test results, treponema pallidum antibody positive, hepatitis B infection (HBsAg or HBcAb positive), hepatitis C infection (HCV antibody positive and quantitative abnormality), cytomegalovirus infection (IgM positive and quantitative abnormality) and Epstein-Barr virus infection (IgM positive and quantitative abnormality);
* 6.History of tuberculosis infection, or evidence of active or latent mycobacterium tuberculosis infection at the time of signing informed consent;
* 7. The following laboratory abnormalities were present, including but not limited to: a) Subjects with abnormal liver function: e.g., aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal (ULN), or total bilirubin > 1.5 × ULN (except for those due to Gilbert syndrome); or b) Subjects with abnormal hematology: Hemoglobin < 90 g/L, or platelet count < 75 x 109/L, or absolute neutrophil count < 1.5 x 109/L;
* 8. Subjects with a history of chronic, recurrent (3 or more infections of the same type within 1 year) or severe infections (e.g. pneumonia and sepsis) within half a year before informed consent as determined by the investigator, including viral infection, or requiring systemic anti-infective treatment within 12 weeks before informed consent;
* 9.History of severe herpes infection (e.g., herpetic encephalitis, ocular herpes or diffuse herpes) or signs of herpes or varicella-zoster virus infection within 12 weeks prior to knowledge (especially chickenpox and herpes zoster);
* 10. History or current history of malignant disease, including solid tumors and hematologic malignancies (except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and cervical cancer in situ that have been completely removed and considered cured > 2 years at the time of informed consent).
* 11. New York Heart Association Functional Class III or IV congestive heart failure
* 12. Subjects with informed consent or abnormal and clinically significant ECG results before administration
* 13.Patients with suicidal behavior or thoughts within 1 year before informed consent;
* 14.Subjects with a history of drug abuse within 12 months before informed consent, or positive baseline urine drug test results;
* 15. Use the prohibited drugs stipulated in the plan
* 16. Antimalarials were started within 12 weeks prior to randomization, and subjects must have been on a stable dose from screening through the end of study (only for CLE patients) if they were receiving antimalarial treatment at screening;
* 17. Treatment with oral systemic corticosteroids at doses greater than 15 mg/day prednisone (or its equivalent) prior to randomization (only for patients with CLE);
* 18. Patients who have previously received drugs that inhibit BDCA2 targets;
* 19. Subjects who have participated in other clinical trials within 4 weeks before informed consent, or within 5 half-lives of the investigational drug, whichever is longer;
* 20. Presence of a past or present condition other than SLE and/or CLE that, in the opinion of the Investigator, may interfere with the assessment of skin inflammation and disease activity;
* 21. Subjects who are allergic to the investigational drug (including excipients) or suffer from serious allergic diseases or have an allergic constitution (such as allergy to two or more drugs, food or pollen), which may impair the safety of subjects in the judgment of the investigator;
* 22. Tattoos, scars or other physical examination findings in the area of planned injection sites that interfere with local injection site evaluation;
* 23. Live vaccine or live attenuated vaccine within 4 weeks before informed consent, or planned during the study and within 24 weeks after the last dose of study drug;
* 24. Subjects with a blood donation volume ≥ 500 mL within 4 weeks before informed consent or planned during the study, or have a history of blood transfusion within 4 weeks before informed consent;
* 25. Subjects with an average daily alcohol intake of more than 2 units (1 unit of alcohol ≈ 360 mL of beer containing 5% alcohol or 45 mL of spirits containing 40% alcohol or 150 mL of wine containing 12% alcohol) within 3 months before informed consent, or subjects with positive baseline alcohol breath test;
* 26. Other reasons that the investigator considers unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-09-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to day 141
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: Results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to 28 Days Post-dose (AUC0-28d) | UP to day 28
Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUClast) | Up to day 141
Cmax of HC022 | Up to day 141
Terminal Elimination Half-Life (t1/2) of HC022 | Up to day 141
Apparent Clearance (CL/F) of HC022 | Up to day 141
Number of Participants Who Develop Serum Anti-HC022 Antibodies | Up to day 141

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China